CLINICAL TRIAL: NCT01410032
Title: Reconstruction Plate Compared With Flexible Intramedullary Nailing for Midshaft Clavicular Fractures: a Prospective, Randomized Clinical Trial
Brief Title: Reconstruction Plate Compared With Flexible Intramedullary Nailing for Midshaft Clavicular Fractures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fernando B Andrade-Silva, MD, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOT-HCFMUSP
Record Dates: First submitted 2011-05-23; First posted 2011-08-04 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Clavicle Fracture
Keywords: clavicle; clavicular; fracture; midshaft; plate; ESIN; intramedullary; flexible; nailing
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plate fixation (Active Comparator): Reconstruction plate
  Interventions: Procedure: Plate fixation
- ESIN (Active Comparator): ESIN (Elastic Stable Intramedullary Nailing)
  Interventions: Procedure: ESIN

INTERVENTIONS:
Procedure: Plate fixation — Reconstruction plate
  Arms: Plate fixation
Procedure: ESIN — ESIN (Elastic Stable Intramedullary Nailing)
  Arms: ESIN

SUMMARY:
The purpose of this study is to compare the clinical and radiographic results of patients with midshaft clavicular fractures treated with plates or intramedullary flexible nails fixation.

DETAILED DESCRIPTION:
Midshaft clavicular fractures are classically treated with non-surgical methods, supported by many authors as an effective treatment. However, different researches have shown high rates of nonunion and clavicle malunion related to the nonoperative treatment. Currently, indications for surgical treatment are wider and include mainly the following: shortening greater than or equal to 2.0 cm, multiple trauma, open fractures or with imminent exposure and associated neurovascular injury.

Plate fixation of midshaft clavicular fractures is widely described in the literature, and is considered the gold standard by different authors, associated with a high union rate and a low complication rate. Different types of plates have been used, including reconstruction plates, dynamic compression plates (DCP), low-contact dynamic compression plates (LC-DCP), semi-tubular plates, and pre-molded locking plates. Possible complications are postoperative infection, hardware loosening or failure, peri-incision paresthesia, neurovascular iatrogenic lesions, nonunion, and hardware related symptoms.

Elastic stable intramedullary nailing (ESIN) technique has been used in recent years in the treatment of midshaft clavicular fractures. Different studies report excellent functional results and low complication rates. Some theoretical advantages in relation to plates are the 3-point flexible nail support, which provides superior biomechanics resistance and uses the relative stability principle, favoring callus formation. When compared to plain steel wires, titanium nails have lower migration risk, due to its greater flexibility and better bone fixation.

The purpose of this study is to compare the clinical and radiographic results of patients with midshaft clavicular fractures treated with reconstruction plates or ESIN.

ELIGIBILITY:
Inclusion Criteria:

1. Displaced Fractures of the middle third of the clavicle (no contact between the main fragments)
2. Age between 16 and 65 year old;
3. Terms of consent signed by the patient or guardian.

Exclusion Criteria:

1. Fracture of medial or lateral third of the clavicle;
2. Cortical contact between the main fracture fragments;
3. Age below 16 years old or more than 65 years old;
4. Pathological fracture;
5. Ipsilateral previous injuries of the shoulder or upper limb;
6. Ipsilateral associated fractures of the shoulder or upper limb;
7. Neuro-vascular injury associated;
8. Open fracture not eligible for primary internal fixation;
9. Clinical contraindication for surgery;
10. Fracture older than 30 days;
11. Patient not cooperative or ineligible for the follow-up;
12. Lack of consent to participate.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-07; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
DASH score | 6 months
  Disabilities of the Arm, Shoulder and Hand score (0: best function; 100: worst function)

SECONDARY OUTCOMES:
DASH score | 12 months
  Disabilities of the Arm, Shoulder and Hand score (0: best function; 100: worst function)
Constant-Murley Score | 6 and 12 months PO
  Shoulder functional score (0: worst function; 100: best function)
Time to Union | Monthly
  Time necessary to reach complete union measured in weeks
Radiographic residual shortening | 6 months
  Clavicles shortening compared to the contralateral side
Patient satisfaction with the treatment | 6 and 12 months
  Subjective measurement. Patients are questioned about their satisfaction with the treatment instituted. Binary outcome.
Complication rate | Monthly
  Complications were divided in Minor and Major, as follows:
  Minor: paresthesia, transient neurologic deficit, implant deformation, partial implant migration, acromioclavicular or sternoclavicular pain, hardware related pain
  Major: permanent neurologic deficit, total implant failure, total implant migration, refracture, reoperation, nonunion

CONTACTS AND LOCATIONS:
Overall Officials: Fernando B Andrade-Silva, MD, Principal Investigator — University of Sao Paulo - Department of Orthopedics and Traumatology
Locations (1):
- University of Sao Paulo - Department of Orthopedics and Traumatology, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Andrade-Silva FB, Kojima KE, Joeris A, Santos Silva J, Mattar R Jr. Single, superiorly placed reconstruction plate compared with flexible intramedullary nailing for midshaft clavicular fractures: a prospective, randomized controlled trial. J Bone Joint Surg Am. 2015 Apr 15;97(8):620-6. doi: 10.2106/JBJS.N.00497. PMID 25878305